CLINICAL TRIAL: NCT01477736
Title: A Comparison Study of Oxybutynin and Botulinum Toxin for Neurogenic Detrusor Overactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Reabilitação e Readaptação Dr. Henrique Santillo (Other)
Responsible Party: Principal Investigator, Ruiter Silva Ferreira, Dr, Centro de Reabilitação e Readaptação Dr. Henrique Santillo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXITBALM
Record Dates: First submitted 2011-11-19; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Spinal Cord Injury
Keywords: Neurogenic bladder; Urodynamic; Quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic | interventions — oxybutynin; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin A (Active Comparator)
  Interventions: Drug: Oxybutynin; Drug: Botulinum toxin A
- oxybutynin (Active Comparator)
  Interventions: Drug: Oxybutynin; Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Oxybutynin — 5 mg of immediate-release oxybutynin orally 3 times daily
Drug: Botulinum toxin A — 300 U intradetrusor injection

SUMMARY:
The purpose of this study is to compare the effects of oral oxybutynin and intradetrusor injections of botulinum toxin type A on urodynamic parameters and quality of life in patients with neurogenic detrusor overactivity following spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* Detrusor overactivity
* Age over 18 years
* Spinal cord injury at least 12 months duration
* Undergoing regular clean intermittent catheterisation

Exclusion Criteria:

* Pregnancy
* Desire to become pregnant during the study period
* Breastfeeding
* Blood coagulation disorder
* Neuromuscular transmission disorder
* Use of any intravesical pharmacologic agents
* Previous use of botulinum toxin A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary study outcome measure was the variation mean in the number of episodes of urinary incontinence per 24 hours, maximum cystometric capacity, maximum detrusor pressure and bladder compliance | Beginning and 24 weeks of the study

SECONDARY OUTCOMES:
The secondary outcome measure was quality of life as measured by the Qualiveen questionnaire | Beginning and 24 weeks of the study

CONTACTS AND LOCATIONS:
Overall Officials: RUITER S FERREIRA, Dr., Principal Investigator — Division of Urology of State University of Campinas, Division of Urology of Centro de Reabilitaçao e Readapatacao Dr. Henrique Santillo
Locations (1):
- UNICAMP, Division of Urology, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Karsenty G, Denys P, Amarenco G, De Seze M, Game X, Haab F, Kerdraon J, Perrouin-Verbe B, Ruffion A, Saussine C, Soler JM, Schurch B, Chartier-Kastler E. Botulinum toxin A (Botox) intradetrusor injections in adults with neurogenic detrusor overactivity/neurogenic overactive bladder: a systematic literature review. Eur Urol. 2008 Feb;53(2):275-87. doi: 10.1016/j.eururo.2007.10.013. Epub 2007 Oct 16. PMID 17988791
- See also: Related Info — http://crer.org.br
- See also: Related Info — http://fcm.unicamp.br